CLINICAL TRIAL: NCT04005092
Title: Helmet Continuous Positive Airway Pressure Versus High Flow Nasal Cannula Oxygen in Acute Cardiogenic Pulmonary Oedema: A Randomized Control Trial
Brief Title: Helmet CPAP Versus HFNC in Acute Cardiogenic Pulmonary Edema
Acronym: HCPAPvsHFNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Raja Permaisuri Bainun (Other Government)
Responsible Party: Principal Investigator, Dr. Adi Bin Osman, EMERGENCY MEDICINE CONSULTANT, Hospital Raja Permaisuri Bainun
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-17-1839-36966
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cardiogenic Pulmonary Edema
Keywords: non invasive ventilation; pulmonary edema; high flow nasal cannula; helmet CPAP; respiratory failure; hyperaemia
MeSH Terms: conditions — Pulmonary Edema; Respiratory Insufficiency; Hyperemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helmet Continuous Positive Airway Pressure(hCPAP) (Active Comparator): Helmet CPAP produce a better physiological outcomes after 1-hour intervention
  Interventions: Device: hCPAP versus HFNC
- High Flow Nasal Cannula(HFNC) (Active Comparator): HFNC produce a better physiological outcomes after 1-hour intervention
  Interventions: Device: hCPAP versus HFNC

INTERVENTIONS:
Device: hCPAP versus HFNC — The patient presented with Acute Cardiogenic Pulmonary Edema will be randomized into either helmet CPAP or HFNC.

SUMMARY:
This study objectively held to compare the physiological outcomes in the non-invasive (NIV) treatment of Acute Cardiogenic Pulmonary Oedema (ACPE) patients in the Emergency Department (ED) delivered by Helmet CPAP (hCPAP) and HFNC.Patients will be randomized to receive either hCPAP or HFNC.

DETAILED DESCRIPTION:
Non-invasive ventilation(NIV) has different types of interfaces that had been used in acute hypoxaemic and hypercapnic respiratory failure. The appropriate interface is necessary to provide comfort and lead to the success of NIV.

Helmet continuous positive airway pressure (hCPAP) is an NIV interface that allows the provision of high airway pressures with a minimal leak.

HFNC which delivers heated humidified high flow oxygen provides a good alternative to the conventional NIV in terms of comfort

ELIGIBILITY:
Inclusion Criteria:

All patients aged more than 18 years old presented with acute cardiogenic pulmonary oedema.

Exclusion Criteria:

1. Age less than 18 years old
2. Low GCS (less than 8), altered mental status
3. Hemodynamic instability, impending cardiopulmonary arrest
4. Use of vasopressors, inotropes
5. Exacerbation of asthma or chronic respiratory failure
6. Urgent need for endotracheal intubation
7. Absence of airway protective gag reflex
8. Elevated intracranial pressure
9. Tracheostomy
10. Pregnant
11. Upper airway obstruction
12. Injuries or surgery to head and neck less than 6 months upon presentation
13. Claustrophobia
14. Blind or poor vision
15. Medico-legal related cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate | 1 hour
  Respiratory rate reduction post intervention

SECONDARY OUTCOMES:
Heart Rate | 1 hour
  Heart rate reduction post intervention
Partial Pressure Of Arterial Oxygen Level | 1 hour
  Partial arterial oxygen level post intervention
Ratio Of Partial Pressure Arterial Oxygen And Fraction Of Oxygen | 1 hour
  Partial arterial oxygen/fraction of oxygen ratio improvement post intervention
Dyspnoea Scale | 1 hour
  Dyspnoea scale improvement post intervention.Dyspnea scale measured using an unmarked 10cm VAS card that had mark with "I can breathe normally", at one end correspond to patients' normal baseline breathing which score "0" and on the other end "I can't breathe at all", which score "10" represent the worst difficulty perceived by patients.
Heart Rate,Acidosis (pH), Consciousness (GCS), Oxygenation (PF ratio) And Respiratory Rate(HACOR) Score | 1 hour
  Heart rate,Acidosis (pH), Consciousness (GCS), Oxygenation (PF ratio) and Respiratory rate(HACOR) Score improvement post intervention.HACOR is an acronym for heart rate, acidosis (pH), consciousness (GCS), oxygenation (PF ratio) and respiratory rate in which each parameter is an independent predictor for NIV failure. HACOR score is out of 25 with differential weighting of each parameter.
Rate Of Intubation | 1 hour
  Intubation rate post intervention
28-Days Mortality In Acute Cardiogenic Pulmonary Edema | 28 days
  Mortality due to Acute Cardiogenic Pulmonary Edema

CONTACTS AND LOCATIONS:
Overall Officials: ADI OSMAN, Principal Investigator — EMERGENCY DEPARTMENT, HOSPITAL RAJA PERMAISURI BAINUN, IPOH, PERAK, MALAYSIA
Locations (1):
- Emergency Department, Hospital Raja Permaisuri Bainun, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osman A, Via G, Sallehuddin RM, Ahmad AH, Fei SK, Azil A, Mojoli F, Fong CP, Tavazzi G. Helmet continuous positive airway pressure vs. high flow nasal cannula oxygen in acute cardiogenic pulmonary oedema: a randomized controlled trial. Eur Heart J Acute Cardiovasc Care. 2021 Dec 18;10(10):1103-1111. doi: 10.1093/ehjacc/zuab078. PMID 34632507

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT04005092/Prot_SAP_000.pdf